CLINICAL TRIAL: NCT04677803
Title: A Phase 2a Multiple Dose Basket Study of the Safety, Tolerability, and Pharmacologic Activity of BT200 in Patients With Hereditary Bleeding Disorders
Brief Title: BT200 in Hereditary Bleeding Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ulla Derhaschnig, MD, Associate Professor, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT200-02
Record Dates: First submitted 2020-12-03; First posted 2020-12-21 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Von Willebrand Diseases; Hemophilia A
MeSH Terms: conditions — von Willebrand Diseases; Hemophilia A

STUDY DESIGN:
Intervention Model Description: Open-label, individual dose titration-to-response, basket trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subcutaneous (SC) injection:
  BT200 dose 3 mg on Day 0, Day 4, and again on Day 7 BT200 dose titrated thereafter between 3 and 9 mg on Days 14, 21, and 28. It is anticipated that dose adjustments will be performed in 2 mg steps. The 9 mg dose will only be applied on day 28 in exceptional circumstances, if no relevant changes in pharmacodynamic and safety parameters will be observed on day 21.
  Interventions: Drug: BT200

INTERVENTIONS:
Drug: BT200 — BT200 is a PEGylated synthetic RNA oligonucleotide

SUMMARY:
BT200 is a PEGylated aptamer that binds to the A1 domain of human von Willebrand factor (VWF). At low doses, BT200 blocks the clearance of VWF antigen (VWF Ag) from the circulation and causes an increase in concentrations of both VWF Ag and Factor VIII (FVIII), but has negligible effect on the activity of either. At higher doses, BT200 blocks clearance of VWF and also inhibits its activity, but still does not inhibit FVIII activity. Therefore, low dose BT200 could potentially be used to correct deficiency of VWF and/or FVIII in patients with hereditary bleeding disorders. This study is designed as a "basket design" pilot study to determine the relevant dose and pharmacological activity of BT200 in such patients.

In this open basket study up to 25 patients with the following congenital blood-clotting disorders are to be included: Patients with hemophilia A, heterozygous carriers of hemophilia A with subnormal FVIII levels; patients with von Willebrand syndrome (VWD) type 1, "Vicenza type", and with VWD type 2b.

Participants will receive BT200 subcutaneously on day 0, day 4 and day 7 in the first week and then once a week for a total of five weeks - initially in a dose of 3 mg, then in week 3 individually after response in a dose of 3 to 9 mg.

Subsequently, blood samples are taken once a week for a further three weeks (wash-out phase).

Patients may be enrolled in an additional pharmacokinetics sub-study. For this purpose, approximately three blood samples are taken to estimate the half-life of substituted FVIII under the influence of BT200.

The primary objective of this study is to obtain clinical proof of mechanism for BT200 in one or more hereditary bleeding disorders.

ELIGIBILITY:
Inclusion Criteria:To be eligible for this study, patients must meet all of the following inclusion criteria:

1. Hereditary bleeding disorder:

   * Congenital hemophilia A without inhibitors with a prophylactic treatment regime
   * Heterozygous carriers of hemophilia A with subnormal FVIII levels
   * VWD Type 1, "Vicenza" type
   * VWD Type 2b
2. Male or female, age ≥18-70 years old at Screening
3. If female, must be post-menopausal or surgically sterilized
4. Able to comprehend and to give informed consent
5. Able to cooperate with the Investigator, to comply with the requirements of the study, and to complete the full sequence of protocol-related procedures -

Exclusion Criteria: Patients meeting any of the following criteria will be excluded from the study:

1. Clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the patient or compromise the quality of the data derived from his/her participation in this study
2. Medical History of spontaneous (not FVIII or FEIBA-associated) venous or arterial thromboembolic events
3. History of significant drug allergy or anaphylactic reactions
4. Substance abuse, mental illness, or any reason that makes it unlikely in the judgment of the Investigator for the patient to be able to comply fully with study procedures
5. Use of medication during 2 weeks before the start of the study, which in the judgment of the Investigator may adversely affect the patient's welfare or the integrity of the study's results
6. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days or 5 elimination half-lives (whichever is longer) prior to treatment start -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Hemophilia A | Baseline through 4 weeks after dosing
  increase in FVIII activity
VWD Type 1 | Baseline through 4 weeks after dosing
  increase in FVIII activity
VWD Type 2b | Baseline through 4 weeks after dosing
  increase in platelet count and/or FVIII activity

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Measured concentration of BT200 (and derived PK parameters) | Baseline through 4 weeks after dosing
  Measured concentration of BT200
Pharmacodynamics | Baseline through 4 weeks after dosing
  PFA-100
Pharmacodynamics | Baseline through 4 weeks after dosing
  Multiplate electrode platelet aggregometer (ristocetin induced)
Pharmacodynamics | Baseline through 4 weeks after dosing
  VWF antigen
Pharmacodynamics | Baseline through 4 weeks after dosing
  VWF:ristocetin co-factor assay
Pharmacodynamics | Baseline through 4 weeks after dosing
  VWF activity
Pharmacodynamics | Baseline through 4 weeks after dosing
  VWF collagen bindign assay
Pharmacodynamics | Baseline through 4 weeks after dosing
  ELISA for unbound VWF-A1 domain
Pharmacodynamics | Baseline through 4 weeks after dosing
  VWF propeptide
Pharmacodynamics | Baseline through 4 weeks after dosing
  Fibrin D-Dimer
Pharmacodynamics | Baseline through 4 weeks after dosing
  Prothrombin fragement (F1.2)
Pharmacodynamics | Baseline through 4 weeks after dosing
  Rotational thrombelastometry
Pharmacodynamics | Baseline through 4 weeks after dosing
  Clot strength assay
Pharmacodynamics | Baseline through 4 weeks after dosing
  Calibrated Thrombogram assay

OTHER OUTCOMES:
Overall safety and tolerability of BT200 | Baseline through 4 weeks after dosing
  Serious, drug-related adverse events (AEs)
Overall safety and tolerability of BT200 | Baseline through 4 weeks after dosing
  Patterns of serious or non-serious, drug-related AEs and/or clinically relevant laboratory abnormalities, vital signs, or physical findings suggestive of one or more specific target organs for toxicity of BT200
Overall safety and tolerability of BT200 | Baseline through 4 weeks after dosing
  Clinically evident bleeding assessed using the International International Society on Thrombosis and Haemostasis (ISTH) Bleeding Score

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Derhaschnig, MD, Principal Investigator — MU Vienna, Dept. of Clinical Pharmacology
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ay C, Kovacevic KD, Kraemmer D, Schoergenhofer C, Gelbenegger G, Firbas C, Quehenberger P, Jilma-Stohlawetz P, Gilbert JC, Zhu S, Beliveau M, Koenig F, Iorio A, Jilma B, Derhaschnig U, Pabinger I. The von Willebrand factor-binding aptamer rondaptivon pegol as a treatment for severe and nonsevere hemophilia A. Blood. 2023 Mar 9;141(10):1147-1158. doi: 10.1182/blood.2022016571. PMID 36108308
- [Derived] Ay C, Pabinger I, Kovacevic KD, Gelbenegger G, Schorgenhofer C, Quehenberger P, Jilma-Stohlawetz P, Sunder-Plassman R, Gilbert JC, Zhu S, Jilma B, Derhaschnig U. The VWF binding aptamer rondoraptivon pegol increases platelet counts and VWF/FVIII in type 2B von Willebrand disease. Blood Adv. 2022 Sep 27;6(18):5467-5476. doi: 10.1182/bloodadvances.2022007805. PMID 35772170